CLINICAL TRIAL: NCT02239237
Title: Post-marketing Safety Surveillance of Compound Kuh-seng Injection: a Registry Study
Status: Completed | Type: Observational
Sponsor: Zhong Wang (Other)
Collaborators: Shanxi Zhendong pharmaceutical Co. LTD. (Unknown)
Responsible Party: Sponsor-Investigator, Zhong Wang, Dr, China Academy of Chinese Medical Sciences
Organization: China Academy of Chinese Medical Sciences (Other)
Other Study IDs: Kuh-seng1.0
Record Dates: First submitted 2014-09-10; First posted 2014-09-12 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Safety Surveillance; Adverse Drug Events; Adverse Drug Reactions; Severe Adverse Events; Severe Adverse Reactions
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum will be retained from the patients who have the anaphylaxis after given the Compound Kuh-seng Injection and the other 4 matched patients who do not has the anaphylaxis.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Compound Kuh-seng Injection: Compound Kuh-seng Injection will be given to the patients, and the investigators will record all the information including ADR, application of Compound Kuh-seng Injection and the combined medications, etc.
  Interventions: Drug: Compound Kuh-seng Injection

INTERVENTIONS:
Drug: Compound Kuh-seng Injection — Compound Kuh-seng Injection is a kind of natural compound injection extracted from Chinese herbs Kuh-seng (Radix Sophorae Flavescentis) and Rhizoma Heterosmilacis Japonicae. The major bioactive ingredients include oxymatrine，sophocarpidine, matrine, flavonoid etc.
  Other Names: Compound Kushen Injection; Fufang Kushen Zhusheye

SUMMARY:
This registry aims to monitor the safety of Compound Kuh-seng Injection and to identify the potential risk factors for the adverse drug reactions. Compound Kuh-seng Injection is a kind of natural compound injection extracted from herbs Kuh-seng (Radix Sophorae Flavescentis) and Rhizoma Heterosmilacis Japonicae.

ELIGIBILITY:
Inclusion Criteria:

* Patients who use Compound Kushen Injection in the monitoring hospitals

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who use Compound Kushen Injection in the monitoring hospitals
Sampling Method: Non-Probability Sample
Enrollment: 30283 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
The incidence of severe adverse reactions (SAR) to the Compound Kuh-seng Injection | 2 years

SECONDARY OUTCOMES:
The incidence of adverse drug reactions (ADR) to Compound Kuh-seng Injection | 2 years
The incidence of anaphylactic reaction to Compound Kuh-seng Injection | 2 years
The incidence of new ADRs to Compound Kuh-seng Injection | 2 years
The incidence of new SARs to Compound Kuh-seng Injection | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Zhong Wang, M.D., Study Director — Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences; Zhan-Yu Pan, Ph.D., Principal Investigator — Tianjin medical university cancer institute & hosptial
Locations (29):
- China (29):
  - HanDan Central Hospital, Handan, Hebei
  - Handan First Hospital, Handan, Hebei
  - Bai Qiu'en International Peace Hospital, Shijiazhuang, Hebei
  - Henan University Huaihe Hospital, Kaifeng, Henan
  - The First Affiliated Hospital of Henan University of Science & Technology, Luoyang, Henan
  - Luoyang Central Hospital Affiliated to Zhengzhou University, Luoyang, Henan
  - Xinxiang Central Hospital, Xinxiang, Henan
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Xinyang Central Hospital, Xinyang, Henan
  - People's Hospital of Zhengzhou, Zhengzhou, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Hospital of Henan College of Traditional Chinese Medicine, Zhengzhou, Henan
  - Shandong Provincial Western Hospital, Jinan, Shandong
  - Qingdao Center Hospital, Qingdao, Shandong
  - Tai'an Central Hospital, Tai’an, Shandong
  - The 88th Hospital of People's Liberation Army, Tai’an, Shandong
  - People's Hospital of Xintai City, Tai’an, Shandong
  - Weifang No.2 People's Hospital, Weifang, Shandong
  - Weihai Municipal Hospital, Weihai, Shandong
  - Central Hospital of Zibo, Zibo, Shandong
  - Jincheng General Hospital, Jincheng, Shanxi
  - The Fourth People's Hospital of Linfen, Linfen, Shanxi
  - Traditional Chinese Hospital of Shanxi, Taiyuan, Shanxi
  - Yuncheng Central Hospital, Yuncheng, Shanxi
  - Chengdu Second People's Hospital, Chengdu, Sichuan
  - AVIC 363 Hospital, Chengdu, Sichuan
  - Teaching Hospital of Chengdu University of T.C.M., Chengdu, Sichuan
  - The Second People's Hospital of Yibin, Yibin, Sichuan
  - Tianjin medical university cancer institute & hosptial, Tianjin, Tianjin Municipality